CLINICAL TRIAL: NCT01527656
Title: Single-Centre, Randomised, Balanced, Double-Blind, Cross-Over Trial Investigating the Bioequivalence of Formulation 2 and Formulation 4 of Biphasic Insulin Aspart 70 in Healthy Male Subjects
Brief Title: Bioequivalence of Two Formulations of Biphasic Insulin Aspart 70 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1577
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- Formulation B (Experimental)
  Interventions: Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 70 — A single dose administrated subcutaneously (s.c., under the skin) on two separate dosing visits. A wash-out period of 6-12 days will take place between dosing visits

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the bioequivalence of two formulations of biphasic insulin aspart 70 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination, as judged by the investigator
* Body Mass Index (BMI) between 19.0-30.0 kg/m^2
* Glycohemoglobin (HbA1c) within laboratory normal range
* Non-smokers

Exclusion Criteria:

* Clinically significant abnormal haematology, biochemistry, urinalysis or ECG (electrocardiogram) screening tests, as judged by the investigator
* Liver enzyme values (ALAT and ASAT) exceeding 2 times the upper reference limit according to the local laboratory
* A history of any illness that, in the opinion of the Investigator and/or Sponsor, might confound the results of the trial or pose additional risk in administering the investigational product to the subject
* History of or current addiction to alcohol or drugs of abuse as determined by the investigator (positive urine drug screen and breath alcohol screen)
* HIV (human immunodeficiency virus), Hepatitis B or C positive
* Subjects with a first-degree relative with diabetes mellitus
* A history of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reactions
* Known or suspected allergy to trial product or related products
* Smoking during the past three months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-12; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart curve in the interval from 0-16 hours
Cmax, maximum insulin aspart concentration

SECONDARY OUTCOMES:
tmax, time to maximum insulin aspart concentration
Area under the insulin aspart curve
Mean residence time (MRT)
t½, terminal half-life
Incidence of hypoglycaemic events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Hanefeld M, Fischer S, Julius U, Schulze J, Schwanebeck U, Schmechel H, Ziegelasch HJ, Lindner J. Risk factors for myocardial infarction and death in newly detected NIDDM: the Diabetes Intervention Study, 11-year follow-up. Diabetologia. 1996 Dec;39(12):1577-83. doi: 10.1007/s001250050617. PMID 8960845
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com